CLINICAL TRIAL: NCT00683254
Title: Analysis of Impact on Nasal Obstruction by Commercially Available Internal Nasal Stents
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator left institution. Project never started.
Sponsor: Bethany L. Jones (Other)
Collaborators: Sanostec Corp. (Industry)
Responsible Party: Sponsor-Investigator, Bethany L. Jones, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: Sanostec-200701751
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Nasal Obstruction
Keywords: nasal obstruction; nasal stent
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Commercially-available internal nasal stents placed inside the nostril should produce decreased nasal obstruction detectable subjectively (volunteers will fill out a survey) and objectively (degree of obstruction will be measured with a rhinomanometer which measure resistant of airflow while breathing through nose).

DETAILED DESCRIPTION:
Nasal rhinomanometry provides a measure of the airflow through the nose during inspiration and expiration. The effect of static obstructions, such as septal deviation, as well as dynamic obstructions, such as lateral nasal wall collapse, can be measured by the rhinomanometer. The effect of commercially available nasal stents on nasal airflow will be measured. In subjects chosen from the general population, some of whom may not complain of nasal obstruction, the airflow will be measured before and after the placement of removable nasal silastic stents. In addition, these subjects will complete a one question scale in the Likert model to rate the degree of their subjective nasal obstruction; they will complete this both before and after placement of the stents. The results of the scale before and after application of the stents will be correlated with the objective measurements of airflow by rhinomanometry taken before and after stent insertion.Several studies have measured the effect of external nasal splints (such as Breathe-Rite strips) on nasal airflow and nasal airway size (as measured by acoustic rhinometry), but few have studied internal nasal stents. No studies have correlated rhinomanometric evaluation of effect on nasal obstruction by nasal stents with the validated NOSE survey (Nasal Obstruction Symptom Evaluation). In patients with a chief complaint of nasal obstruction and who are noted to have anterior nasal obstruction, nasal stents may provide a satisfactory improvement in nasal airflow without surgical or medicinal intervention. For patients who are determined to be candidates for surgical intervention, the surgical procedure is tailored to their specific anatomic deformities, as determined by the staff facial plastic surgeon. While the patient's complaint of nasal obstruction as well as the surgeon's assessment of the nasal anatomy are important components in the determination of the need for surgical intervention, no studies have utilized the validated NOSE instrument of subjective complaint of nasal obstruction combined with objective measurements of dynamic airflow. Rhinomanometric measurements can be used to further validate the NOSE instrument both preoperatively and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older

Exclusion Criteria:

* history of nasal surgery, currently using topical nasal steroid spray, over the counter decongestant, history of recurrent epistaxis or history of nosebleed within 2 weeks prior to data collection, currently pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our subject pool will be comprised of healthy volunteers, at least 18 years of age, who have not had nasal surgery, are not currently using a topical decongestant, topical nasal steroid spray, or over the counter decongestant, and have no history of recurrent epistaxis or a running nosebleed within 2 weeks prior to data collection.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2008-08 (Estimated); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
change in resistance to airflow after stents inserted as measured by rhinomanometer | data collection occurs at one time only, takes less than 5 minutes to record

SECONDARY OUTCOMES:
subjective decrease in nasal obstruction after stents placed recorded by volunteers filling out a survey | recorded at time of stent placement, one time only

CONTACTS AND LOCATIONS:
Overall Officials: Bethany L Jones, MD, Principal Investigator — University of Iowa Department of Otolaryngology; Grant Hamilton, MD, Study Director — University of Iowa Department of Otolaryngology
Locations (1):
- University of Iowa Department of Otolaryngology, Iowa City, Iowa, United States

REFERENCES:
- [Background] Lam DJ, James KT, Weaver EM. Comparison of anatomic, physiological, and subjective measures of the nasal airway. Am J Rhinol. 2006 Sep-Oct;20(5):463-70. doi: 10.2500/ajr.2006.20.2940. PMID 17063739
- [Background] Wong LS, Johnson AT. Decrease of resistance to air flow with nasal strips as measured with the airflow perturbation device. Biomed Eng Online. 2004 Oct 22;3(1):38. doi: 10.1186/1475-925X-3-38. PMID 15500689
- [Background] Suzina AH, Hamzah M, Samsudin AR. Objective assessment of nasal resistance in patients with nasal disease. J Laryngol Otol. 2003 Aug;117(8):609-13. doi: 10.1258/002221503768199933. PMID 12956914
- [Background] Huang TW, Cheng PW. Changes in nasal resistance and quality of life after endoscopic microdebrider-assisted inferior turbinoplasty in patients with perennial allergic rhinitis. Arch Otolaryngol Head Neck Surg. 2006 Sep;132(9):990-3. doi: 10.1001/archotol.132.9.990. PMID 16982976